CLINICAL TRIAL: NCT00672919
Title: A Single-Arm, Open-Label, Multicenter Study Evaluating the Triglyceride Changes in Subjects With Type 2 Diabetes Mellitus and Dyslipidemia Following Treatment Conversion From Rosiglitazone to Pioglitazone HCl in Combination With Stable Statin Therapy
Brief Title: Pioglitazone Study of Triglyceride Changes in Subjects With Type 2 Diabetes After Conversion From Rosiglitazone.
Acronym: COMPLEMENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-03-TL-OPI-523; U1111-1115-8914 (Registry Identifier: WHO)
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pioglitazone QD (Experimental): (and stable statin therapy)
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone 30 mg to 45 mg, tablets, orally, once daily in combination with stable statin therapy for up to 17 weeks.
  Other Names: ACTOS®; AD-4833

SUMMARY:
The purpose of this study is to measure the triglyceride changes in subjects with type 2 diabetes mellitus taking pioglitazone, once daily (QD), following treatment conversion from rosiglitazone.

DETAILED DESCRIPTION:
Diabetes mellitus is a chronic disease with multiple metabolic defects that result in hyperglycemia arising from inadequate insulin activity. Type 2 diabetes has a genetic predisposition, but lifestyle, physical habits and age play important roles in determining its time of onset and severity. Type 2 diabetes is usually the result of a progression from reduced sensitivity of hepatic (liver) and peripheral-tissue cells to circulating insulin (ie, insulin resistance) to a progressive inability of the body to produce adequate insulin to overcome insulin resistance (ie, insulin deficiency due to beta-cell insufficiency) resulting in impaired glucose tolerance and ultimately overt diabetes. In the United States, an estimated 15.7 million people have diabetes, with type 2 diabetes occurring in approximately 90 to 95% of cases.

Therapeutic agents have been developed to address each of the major functional metabolic defects associated with type 2 diabetes. Recently introduced drugs for diabetes therapy are the thiazolidinedione class. Thiazolidinediones increase glucose utilization, decrease gluconeogenesis and increase glucose disposal through an incompletely understood mechanism but one associated with binding of the drug to receptors known as peroxisomal proliferator-activated receptors.

Thiazolidinediones are peroxisomal proliferator-activated receptor agonists reducing insulin resistance in muscle cells, adipose (fat) tissue, and hepatic cells (inhibiting hepatic gluconeogenesis) with no direct impact on insulin secretion. Thus peroxisomal proliferator-activated receptor agonists improve glycemic control and result in reduced levels of circulating insulin. Peroxisomal proliferator-activated receptors are found in various tissues important for insulin action, with the greatest concentration of these receptors is in adipose tissue.

Pioglitazone is a peroxisomal proliferator-activated receptor agonist developed by Takeda Chemical Industries, Ltd. (Osaka, Japan).

Participation in this study is anticipated to be approximately 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study
* Has been taking a stable dose of rosiglitazone for greater than 90 days prior to screening.
* Has a triglyceride level greater than 200 mg per dL but less than 1000 mg per dL.
* Has been taking a stable statin therapy for greater than 90 days prior to screening.
* Has a glycosylated hemoglobin less than 10.5%.

Exclusion Criteria:

* Type 1 diabetes mellitus.
* Treated with Gemfibrozil within 90 days of screening.
* Previous history of cancer, other than basal cell carcinoma, that has not been in remission for at least 5 years prior to the first dose of study drug.
* The subject has an alanine aminotransaminase level of greater than 2.5 times the upper limit of normal, active liver disease, or jaundice.
* Male subjects who have serum creatinine greater than 2.0 mg per dL and female subjects with serum creatinine greater than1.8 mg per dL.
* Unexplained microscopic hematuria greater than plus 1 confirmed by repeat testing.
* Male subjects who have hemoglobin less than 10.5 g per dL and female subjects who have hemoglobin less than 10.0 g per dL.
* Significant cardiovascular disease including, but not limited to, New York Heart Association Functional (Cardiac) Classification III or IV
* Currently is participating in another investigational study or has participated in an investigational study within the past 30 days.
* Any other serious disease or condition that might affect life expectancy or make it difficult to successfully manage and follow the subject according to the protocol.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Glucocorticoids (eg. prednisone, cortisone, hydrocortisone, dexamethasone) with the exception of a topical glucocorticoid agent.
  * Gemfibrozil
  * Steroid-joint injections.
  * Thiazolidinediones with the exception of the study medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2003-11; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Triglyceride Levels | Weeks 8 and 17 or Final Visit

SECONDARY OUTCOMES:
Change from Baseline in Total Cholesterol | Weeks 8 and 17 or Final Visit
Change from Baseline in direct Low Density Lipoprotein cholesterol | Weeks 8 and 17 or Final Visit
Change from Baseline in High Density Lipoprotein cholesterol | Weeks 8 and 17 or Final Visit
Change from Baseline in apolipoprotein B (apoB) | Weeks 8 and 17 or Final Visit
Change from Baseline in apolipoprotein A1 (apoA1) | Weeks 8 and 17 or Final Visit
Change from Baseline in Free Fatty Acids | Weeks 8 and 17 or Final Visit
Change from Baseline in Lipid Fractionation | Weeks 8 and 17 or Final Visit
Change from Baseline in C-reactive Protein | Weeks 8 and 17 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science Strategy, Study Director — Takeda
Locations (53):
- United States (51):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Bellflower, California
  - Burlingame, California
  - Fresno, California
  - La Jolla, California
  - Long Beach, California
  - Pasadena, California
  - Arvada, Colorado
  - Norwalk, Connecticut
  - Waterbury, Connecticut
  - Aventura, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - North Miami Beach, Florida
  - Tallahassee, Florida
  - West Palm Beach, Florida
  - Columbus, Georgia
  - Idaho Falls, Idaho
  - Chicago Heights, Illinois
  - Evansville, Indiana
  - Des Moines, Iowa
  - Lafayette, Louisiana
  - Fall River, Massachusetts
  - Waltham, Massachusetts
  - Tupelo, Mississippi
  - Chesterfield, Missouri
  - Omaha, Nebraska
  - Staten Island, New York
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Centerville, Ohio
  - Dayton, Ohio
  - Medford, Oregon
  - Meadville, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Warwick, Rhode Island
  - Chattanooga, Tennessee
  - Morristown, Tennessee
  - Murfreesboro, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Houston, Texas
  - Midland, Texas
  - San Antonio, Texas
  - Ogden, Utah
  - Orange, Virginia
  - Virginia Beach, Virginia
  - Man, West Virginia
  - Wausau, Wisconsin
- Puerto Rico (2):
  - Carolina
  - Ponce

REFERENCES:
- [Background] Berhanu P, Kipnes MS, Khan MA, Perez AT, Kupfer SF, Spanheimer RC, Demissie S, Fleck PR. Effects of pioglitazone on lipid and lipoprotein profiles in patients with type 2 diabetes and dyslipidaemia after treatment conversion from rosiglitazone while continuing stable statin therapy. Diab Vasc Dis Res. 2006 May;3(1):39-44. doi: 10.3132/dvdr.2006.005. PMID 16784180
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI